CLINICAL TRIAL: NCT05962294
Title: The Efficacy and Safety of Oxycodone Hydrochloride Sustained-release Tablets in the Treatment of Moderate to Severe Cancer Pain：A Multicenter Real World Study
Brief Title: Real World Study of Oxycodone Sustained-release Tablets for Patients With Moderate to Severe Cancer Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: TA2023-246
Record Dates: First submitted 2023-07-06; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Cancer Pain; Real-world Study; Oxycodone
Keywords: Oxycodone Hydrochloride Sustained-release Tablets
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this real world study is to observe the efficacy and safety of Oxycodone Hydrochloride Sustained-release Tablets in the treatment of moderate to severe cancer pain participants in real clinical practice.

After entering the study, participants will take Oxycodone Hydrochloride Sustained-release Tablets. The investigators need to observe and record relevant data, and finally analyze and summarize the data to understand the efficacy and safety.

DETAILED DESCRIPTION:
This study is a prospective, single arm, multicenter real world study, the investigators didn't set up a control group. After the participant is enrolled, the participant will enter a 14 day treatment cycle, where the medication will be proportionally converted into Oxycodone Hydrochloride Sustained-release Tablets. The daily medication dose will be adjusted based on the number of pain outbreaks and pain scores (According to the drug increment principle of NCCN), and various information (Daily oxycodone dose, average pain score, minimal pain score, most severe pain score, number of breakout pain, name of rescue drugs, number of rescue, heart rate, blood pressure, respiratory rate, SPO2, combination of drugs, pain control satisfaction, etc) about the participant's medication will be recorded. The participant will not be limited to whether to combine medication. Observe the efficacy and safety of Oxycodone Hydrochloride Sustained-release Tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an informed consent form;
2. Age ≥ 18 years old;
3. Patients with moderate to severe (NRS ≥ 4 points) cancer pain;
4. Patients with oral equivalent Oxycodone Hydrochloride Sustained-release Tablets ≥ 80mg/d.

Exclusion Criteria:

1. Patients with severe mental illness who cannot cooperate with follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a prospective, single arm, multicenter real-world study that only needs to meet the requirements of age, disease type, drug dosage, and no severe mental illness in the study population
Sampling Method: Non-Probability Sample
Enrollment: 916 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Mean difference in pain intensity after treatment | From the 1st to 14th day of treatment
  Use the Numeric Rating Scale（NRS, 0 to 10 points, lower scores indicate better pain control） to evaluate the average pain score per day over the past 24 hours. Calculate the daily difference in pain intensity (PID) by subtracting the daily NRS score from the baseline NRS score. Divide the sum of PID on days 1 to 14 by 14 to obtain the mean difference in pain intensity (MPID).
The proportion of patients with effective pain relief | From the 1st to 14th day of treatment
  Effective pain relief is defined as a decrease of 30% or more in average pain intensity from day 1 to day 14 compared to the baseline period.

SECONDARY OUTCOMES:
The proportion of patients with effective pain control | From the 1st to 14th day of treatment
  The proportion of patients whose pain is under control. It requires the Numeric Rating Scale (NRS, 0 to 10 points, lower scores indicate better pain control) is ≤ 3 points, and the break-through cancer pain is ≤ 3 times per day.
The time for the patient's pain to be effectively controlled | From the 1st to 14th day of treatment
  The time from the beginning of treatment to effective pain control for patients. It requires the Numeric Rating Scale (NRS, 0 to 10 points, lower scores indicate better pain control) is ≤ 3 points, and the break-through cancer pain is ≤ 3 times per day.
The improvement of patient symptoms | On the 3rd, 7th, and 14th days after treatment
  We use the Brief Pain Inventory (BPI) to evaluate the improvement of patient symptoms. There are a total of 7 projects, with each project scoring 0-10 points. The lower the score, the more significant the improvement in symptoms.
The satisfaction with pain control | On the 3rd, 7th, and 14th days after treatment
  0-10 points (the higher the score, the higher the satisfaction), participants can rate treatment satisfaction based on the efficacy and safety of the experimental drug. It's the patient's subjective perception of pain control.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China